CLINICAL TRIAL: NCT04516161
Title: Patients With Metastatic Castrate-resistant Prostate Cancer (mCRPC) Treated With Radium-223 (Xofigo): Patient Characteristics and Predictors of Long-term Survival
Brief Title: EPIX, a Study to Gather More Information About Characteristics of Patients and Other Factors Which May Contribute to Survival Over a Long Period of Time in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC) Treated With Radium-223 (Xofigo)
Acronym: EPIX
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20977
Record Dates: First submitted 2020-07-27; First posted 2020-08-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223 dichloride (Xofigo, BAY88-8223): Patients with mCRPC who received treatment of Ra-223.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Receiving Ra-223 either alone or in combination with other cancer therapies at any time after diagnosis of mCRPC

SUMMARY:
In this observational study researchers want to gather more information about the characteristics of patients treated with Radium-223 (Xofigo) who had survived over a long period of time prostate cancer that had spread to other places in the body and keeps growing even when the amount of testosterone in the body is reduced to very low levels (metastatic castration-resistant prostate cancer, mCRPC). In addition researchers want to identify the factors which may contribute to survival over a long period of time in those patients. Radium-223 (Ra-223) is an alpha particle-emitting radioactive agent approved for the treatment of men with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion criteria

* Adult patients with documented diagnosis of mCRPC (≥18 years at diagnosis), and
* Received Ra-223 as one of the therapies between Jan 1, 2013 and Jun 31, 2019 after diagnosis of mCRPC

Exclusion criteria

- Patients involved in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRPC who received Ra-223 from the Bayer Flatiron Xofigo Registry database (BFXR, Version Mar, 2020 with a data cutoff date of Dec, 2019). The database currently includes 1,372 patients with mCRPC who received Ra-223.
Sampling Method: Non-Probability Sample
Enrollment: 1180 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Overall survival from initiation of Ra-223 | Retrospective analysis from Jan 2013 to Dec 2019

SECONDARY OUTCOMES:
Percentage of Prostate Specific Antigen (PSA) (unit: µg/L) response after Ra-223 | Retrospective analysis from Jan 2013 to Dec 2019
  PSA response will be defined ≥ 50% reduction in baseline PSA level after initiation of Ra-223

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer Flatiron Xofigo Registry database, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] George DJ, Agarwal N, Sartor O, Sternberg CN, Tombal B, Saad F, Miller K, Constantinovici N, Guo H, Reeves J, Jiao X, Sandstrom P, Verholen F, Higano CS, Shore N. Real-world patient characteristics associated with survival of 2 years or more after radium-223 treatment for metastatic castration-resistant prostate cancer (EPIX study). Prostate Cancer Prostatic Dis. 2022 Feb;25(2):306-313. doi: 10.1038/s41391-021-00488-0. Epub 2022 Feb 21. PMID 35190653